CLINICAL TRIAL: NCT02818842
Title: Evaluation of Drug's Risk in Pregnant Women
Acronym: EFEMERIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/16-7917
Record Dates: First submitted 2016-06-23; First posted 2016-06-30 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy
Keywords: Database; Birth defects; Neonatal pathologies
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Medical and personal data will be collected for all the pregnant women who want to participate.
  The source of data are :
  * Primary Health Insurance Fund data
  * Prenatal Diagnostic Center of Toulouse University Hospital data
  * Mother and child protection data collection
  * Medicalisation Program of Information Systems data
  Interventions: Other: Primary Health Insurance Fund data; Other: Prenatal Diagnostic Center of Toulouse University Hospital data; Other: Mother and child protection data collection; Other: Medicalisation Program of Information Systems data

INTERVENTIONS:
Other: Primary Health Insurance Fund data — Data collected are:
  * First and last name of mother
  * Age
  * Mother's date of birth
  * Theorical date of beginning of pregnancy
  * Childbirth date
Other: Prenatal Diagnostic Center of Toulouse University Hospital data — Data collected are :
  * First and last name of the mother
  * Mother's birth date
  * Mother Obstetric history
  * Course of pregnancy
  * Drug exposure (name, decision period)
  * Medical termination of pregnancy (date, cause ...)
  * Malformations (description, test results, gender of the child,
  * Weight, height and head circumference, American Pediatric Gross Assessment Record, neonatal pathology).
Other: Mother and child protection data collection — Date collected are :
  * Name and surname of Mother
  * Date of birth of the mother
  * Obstetric history of the mother (the first certificate to 8 days)
  * Course of pregnancy (1st certificate to 8 days)
  * Birth data (1 certificate to 8 days)
  * Child gender,
  * Age of the child at the time of the review,
  * Weight, height and head circumference of the child
  * American Pediatric Gross Assessment Record (1 certificate to 8 days)
  * Neonatal diseases (1 certificate to 8 days)
  * Birth defects (1 certificate to 8 days)
  * Death (age at death)
  * History (certificates at 9 and 24 months)
  * Current diseases (certificates at 9 and 24 months)
  * Psychomotor development (certificates at 9 and 24 months).
  * Date of drugs issue
  * Amount of drug issued
  * Type of feeding (1 certificate to 8 days)
Other: Medicalisation Program of Information Systems data — Data collected are :
  * First and last name of the mother
  * Mother's birth date
  * History of abortions (date and cause)

SUMMARY:
Medication during pregnancy can lead to the occurrence of birth defects or neonatal pathologies. Thalidomide or diethylstilbestrol (Distilbene°) are prominent examples. Many drugs remain insufficiently evaluated in this area and doctors are too often deprived of relevant information when prescribing drugs in pregnant women.

DETAILED DESCRIPTION:
To fill this gap, the investigators have put in place since 2004, a database, EFEMERIS, recording products given to women during pregnancy in Haute-Garonne (data from Primary Health Insurance Fund), fate of these pregnancies and the state health of newborns (Mother and child protection data, prenatal Diagnostic Centre and Medicalisation Program of Information Systems data).

Women included in this database (> 90 000 to date) has allowed us to study the risks of taking certain medications still not assessed in pregnant women (for example phloroglucinol, the H1N1 flu vaccine , oseltamivir ...). Each year about 10 000 pregnant women join the cohort. The collection and management of data concerning require careful organization and mobilize multiple stakeholders.

The pursuit of these inclusions is needed to study medication less often prescribed but raise questions. For example, if the investigators consider that the relative risk of cardiac abnormalities following in utero exposure to paroxetine is multiplied by 1.5, it will take 1,000 women exposed to paroxetine for 5 additional cases observed. In December 2013, 0.3% of women EFEMERIS were exposed to paroxetine in the first quarter (274 women).

The objective of this project is to continue the EFEMERIS project (funded for 10 years public tenders until December 2015) by continuing to include pregnant women (about 10 000 per year) in order to explore the potential effects of exposure to different drugs on the newborn (prematurity, birth defects, neonatal diseases).

The processing of data will EFEMERIS to detect drugs at risk to the fetus and provide a warning role in terms of malformation effects, to monitor over time prescribing practices, participate in pharmacoepidemiology international multicenter studies including similar databases in general population.

ELIGIBILITY:
Inclusion Criteria:

* Women supported by the general scheme of the Primary Health Insurance Fund of the Haute-Garonne who gave birth or had a miscarriage between 1 January 2015 and 31 december 2017.
* Women not opposing that us to access to their data.
* Women for which at least one baby health certificate has been registered at the Mother and child protection, or the outcome of pregnancy was identified by prenatal diagnosis center or Medicalisation Program of Information Systems.

Exclusion Criteria:

* Women that refuses to give access to the data concerning them.
* Women for which no data on pregnancy outcome can be collected.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes women supported by the general scheme of the Primary Health Insurance Fund of the Haute-Garonne in the framework of maternity insurance.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of risk to drug exposition in utero as assessed by descriptive analysis of data gathered | Through the study completion, an average of 36 months
  Analysis of all data collected from the four sources of information :
  * Primary Health Insurance Fund
  * Medicalisation Program of Information Systems
  * Mother and child protection
  * Prenatal Diagnostic Center of Toulouse University Hospital

SECONDARY OUTCOMES:
Assessment of risk associated with non prescription drugs during pregnancy as assessed by descriptive analysis of data gathered | Through the study completion, an average of 36 months
  Analysis of all data collected from the four sources of information :
  * Primary Health Insurance Fund
  * Medicalisation Program of Information Systems
  * Mother and child protection
  * Prenatal Diagnostic Center of Toulouse University Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christine Damase-Michel, PHD, Study Director — University of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hurault-Delarue C, Lacroix I, Benard-Laribiere A, Montastruc JL, Pariente A, Damase-Michel C. Antidepressants during pregnancy: a French drug utilisation study in EFEMERIS cohort. Eur Arch Psychiatry Clin Neurosci. 2019 Oct;269(7):841-849. doi: 10.1007/s00406-018-0906-2. Epub 2018 May 26. PMID 29804133